CLINICAL TRIAL: NCT02634333
Title: Intravitreous Anti-Vascular Endothelial Growth Factor Treatment for Prevention of Vision Threatening Diabetic Retinopathy in Eyes at High Risk
Brief Title: Anti-VEGF Treatment for Prevention of PDR/DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Juvenile Diabetes Research Foundation (Other); National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DRCR.net Protocol W; EY14231 (Other Grant/Funding Number: National Eye Institute); EY23207 (Other Grant/Funding Number: National Eye Institute); EY18817 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2015-12-11; First posted 2015-12-18 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: anti-vascular endothelial growth factor; nonproliferative diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (Prompt Sham) (Sham Comparator): Sham injection in study eye at randomization and at visits at 1, 2, and 4 months and then every 4 months thereafter. Deferred aflibercept may be given if center-involved diabetic macular edema or proliferative diabetic retinopathy develops and deferred laser may subsequently be added to intravitreal aflibercept if certain criteria are met.
  Interventions: Procedure: Prompt Sham; Procedure: Deferred laser; Drug: Deferred aflibercept
- Prompt aflibercept (Experimental): Aflibercept injection in study eye at randomization and at visits at 1, 2, and 4 months and then every 4 months thereafter. More frequent aflibercept may be given if center-involved diabetic macular edema or proliferative diabetic retinopathy develops and deferred laser may subsequently be added to intravitreal aflibercept if certain criteria are met.
  Interventions: Drug: Prompt aflibercept; Procedure: Deferred laser; Drug: Deferred aflibercept

INTERVENTIONS:
Procedure: Prompt Sham — A sham injection (syringe without a needle pressed against the injection site) is performed on the day of randomization and visits at 1, 2, and 4 months and then every 4 months thereafter.
  Arms: Observation (Prompt Sham)
Drug: Prompt aflibercept — Intravitreal injection of 2.0mg aflibercept is performed on the day of randomization and visits at 1, 2, and 4 months and then every 4 months thereafter.
  Other Names: intravitreal anti-vascular endothelial growth factor; Eylea
  Arms: Prompt aflibercept
Procedure: Deferred laser — Laser (either focal/grid laser for diabetic macular edema or panretinal photocoagulation for proliferative diabetic retinopathy) is added following initiation of anti-vascular endothelial growth factor injections for center-involved diabetic macular edema or proliferative diabetic retinopathy only if certain criteria are met
  Other Names: focal/grid photocoagulation; panretinal photocoagulation
Drug: Deferred aflibercept — Intravitreal injection of 2.0mg aflibercept performed once proliferative diabetic retinopathy or center-involved diabetic macular edema develops and then up to every 4 weeks using defined treatment criteria.
  Other Names: intravitreal anti-vascular endothelial growth factor; Eylea

SUMMARY:
Multiple studies have implicated vascular endothelial growth factor VEGF as a major causative factor in human eye diseases characterized by neovascularization including proliferative diabetic retinopathy (PDR) and vascular permeability including diabetic macular edema (DME). While there is strong evidence that PDR outcomes are markedly reduced in eyes that are treated with monthly anti-VEGF therapy (A Study of Ranibizumab Injection in Subjects With Clinically Significant Macular Edema (ME) With Center Involvement Secondary to Diabetes Mellitus: RIDE/RISE) and moderately reduced in eyes that received fairly frequent dosing during the 1st year of treatment (Diabetic Retinopathy Clinical Research Network protocol I), it is unknown whether or not an earlier but less frequent dosing regimen would result in similar, favorable anatomic outcomes, and whether favorable anatomic outcomes subsequently would result in favorable visual acuity outcomes.

If this study demonstrates that intravitreous aflibercept treatment is effective and safe for reducing the onset of PDR or center involved- DME (CI-DME) in eyes that are at high risk for these complications, a new strategy to prevent vision threatening complications of diabetes will be available for patients. The application of intravitreous aflibercept earlier in the course of disease (i.e., at the time when an eye has baseline severe non-proliferative diabetic retinopathy) could help to reduce future potential treatment burden in patients, at the same time resulting in similar or better long-term visual outcomes, if PDR and DME are prevented.

The primary objectives of this protocol are to 1) determine the efficacy and safety of intravitreous aflibercept injections versus sham injections (observation) for prevention of PDR or CI-DME in eyes at high risk for development of these complications and 2) compare long-term visual outcomes in eyes that receive anti-VEGF therapy early in the course of disease with those that are observed initially, and treated only if high-risk PDR or CI-DME with vision loss develops.

Secondary objectives include:

* Comparing other visual acuity outcomes between treatment groups, such as proportion of eyes with at least 10 or at least 15 letter loss from baseline, or gain or loss of at least 5 letters at the consecutive study visit just before and at the 2- or 4-year visit
* Comparing optical coherence tomography (OCT) outcomes, such as mean change in OCT central subfield thickness and volume from baseline
* Comparing proportion of eyes with at least 2 and 3-step worsening or improvement of diabetic retinopathy severity level (scale for individual eyes) by central reading center from baseline
* Comparing associated treatment and follow-up exam costs between treatment groups
* Comparing safety outcomes between treatment groups

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   • Any one of the following will be considered to be sufficient evidence that diabetes is present:
   1. Current regular use of insulin for the treatment of diabetes
   2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   3. Documented diabetes by American Diabetes Association and/or World Health Organization criteria
3. Able and willing to provide informed consent.

Meets all of the following ocular criteria in at least one eye:

1. Best corrected Electronic-Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity letter score ≥79 (approximate Snellen equivalent 20/25 or better)
2. Severe non-proliferative diabetic retinopathy (NPDR) (based on the 4:2:1 rule) evident on clinical examination and on digital imaging as judged by the investigator. Reading center grading of less than ETDRS level 43 or greater than 53 is an exclusion.

   Severe NPDR is defined as:
   1. All 4 midperipheral quadrants show severe hemorrhages or microaneurysms (at least as great as Standard photograph 2A, approximately 20 dot and blot hemorrhages), or
   2. At least 2 fields of definite venous beading in the midperipheral quadrants or at least 1 field at least as severe as Standard photograph 6A, or
   3. At least 1 field of moderate intraretinal microvascular abnormalities (IRMA) in the midperipheral quadrants, at least as severe as Standard photograph 8A
3. No evidence of neovascularization on clinical exam including active neovascularization of the iris (small iris tufts are not an exclusion) or angle neovascularization (if the angle is assessed).
4. No evidence of neovascularization (NV) on fluorescein angiography within the 7-modified ETDRS fields, confirmed by the central Reading Center prior to randomization.

   • The widest method of imaging available at the site must be used to document whether there is NV present in the periphery; however, presence of NV outside of the 7-modified ETDRS fields on ultrawide field imaging will not be an exclusion provided treatment is not planned.
5. No center-involved diabetic macular edema (CI-DME) on clinical exam and optical coherence tomography (OCT) central subfield thickness must be below the following gender and OCT-machine specific thresholds:

   1. Zeiss Cirrus: 290 µm in women and 305 µm in men
   2. Heidelberg Spectralis: 305 µm in women and 320 µm in men
   3. Investigator and potential participant are comfortable withholding treatment for DME until there is at least a 10% increase in OCT central subfield thickness with confirmed visual acuity loss (10 letter loss at a single visit or 5 to 9 at two consecutive visits).
6. Prompt panretinal photocoagulation (PRP) or anti-vascular endothelial growth factor (anti-VEGF) treatment not required AND investigator and potential participant are willing to wait for development of high-risk characteristics (defined in protocol) to treat PDR.
7. Media clarity, pupillary dilation, and study participant cooperation sufficient to obtain adequate fundus photographs, fluorescein angiogram, and OCT.

   * Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality (including segmentation line placement)

Exclusion Criteria:

1. History of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months.
4. Participation in an investigational trial that involved treatment within 30 days of randomization with any drug that has not received regulatory approval for the indication being studied.

   • Note: study participants cannot participate in another investigational trial that involves treatment with an investigational drug while participating in the study.
5. Known allergy to any component of the study drug or any drug used in the injection prep (including povidone iodine prep).
6. Known allergy to fluorescein dye.
7. Blood pressure > 180/110 (systolic above 180 or diastolic above 110). • If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
8. Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.

   • These drugs should not be used during the study.
9. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 2 years.

   • Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
10. Individual is expecting to move out of the area of the clinical center to an area not covered by another Diabetic Retinopathy Clinical Research Network certified clinical center during the next 2 years.

Individual has any of the following ocular characteristics in the eye(s) being evaluated:

1. Exam or photographic evidence of vitreous hemorrhage or preretinal hemorrhage presumed to be from PDR.
2. History of prior vitreous hemorrhage or preretinal hemorrhage presumed to be from PDR.
3. History of prior PRP (defined as ≥100 burns outside of the posterior pole).
4. An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, vitreomacular traction, etc.).
5. History of DME or diabetic retinopathy treatment with laser or intraocular injections of medication within the prior 12 months and no more than 4 prior intraocular injections at any time in the past.

   • Enrollment will be limited to a maximum of 25% of the planned sample size with any history of treatment for DME and/or diabetic retinopathy. Once this number of eyes has been enrolled, any history of treatment for DME and/or diabetic retinopathy will be an exclusion criterion.
6. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
7. Any history of vitrectomy.
8. History of yttrium aluminum garnet capsulotomy performed within 2 months prior to randomization.
9. Aphakia.
10. Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis.
11. Evidence of uncontrolled glaucoma.

    * Intraocular pressure must be <30, with no more than one topical glaucoma medication, and no documented glaucomatous field loss for the eye to be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K. Sun, MD, MPH, Study Chair — Joslin Diabetes Center
Locations (85):
- United States (81):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - University of Arizona Medical Center/Department of Ophthalmology, Tucson, Arizona
  - Atlantis Eye Care, Huntington Beach, California
  - Loma Linda University Health Care, Department of Ophthalmology, Loma Linda, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Southern California Desert Retina Consultants, MC, Palm Desert, California
  - Shashi D Ganti, MD PC, Porterville, California
  - Retina Consultants of Southern California, Redlands, California
  - U.C. Davis Eye Center, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - New England Retina Associates, Hamden, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville Health Science Cent, Jacksonville, Florida
  - Florida Retina Institute-Jacksonville, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Florida Retina Institute, Orlando, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, P.A., Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - Mid-America Retina Consultants, P.A., Kansas City, Missouri
  - Retinal and Ophthalmic Consultants, PC, Northfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - MaculaCare, New York, New York
  - University of Rochester, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Western Carolina Clinical Research, LLC, Asheville, North Carolina
  - Kittner Eye Center, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Carolina Retina Center, Columbia, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Robert E. Torti, MD, PA dba Retina Specialists, DeSoto, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Dept. of Ophthalmology, Richmond, Virginia
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
- Canada (4):
  - UBC/VCHA Eye Care Centre, Vancouver, British Columbia
  - Nova Scotia District Health Authority, Halifax, Nova Scotia
  - Toronto Retina Institute (TRI), North York, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Maturi RK, Glassman AR, Josic K, Baker CW, Gerstenblith AT, Jampol LM, Meleth A, Martin DF, Melia M, Punjabi OS, Rofagha S, Salehi-Had H, Stockdale CR, Sun JK; DRCR Retina Network. Four-Year Visual Outcomes in the Protocol W Randomized Trial of Intravitreous Aflibercept for Prevention of Vision-Threatening Complications of Diabetic Retinopathy. JAMA. 2023 Feb 7;329(5):376-385. doi: 10.1001/jama.2022.25029. PMID 36749332
- [Derived] Maturi RK, Glassman AR, Josic K, Antoszyk AN, Blodi BA, Jampol LM, Marcus DM, Martin DF, Melia M, Salehi-Had H, Stockdale CR, Punjabi OS, Sun JK; DRCR Retina Network. Effect of Intravitreous Anti-Vascular Endothelial Growth Factor vs Sham Treatment for Prevention of Vision-Threatening Complications of Diabetic Retinopathy: The Protocol W Randomized Clinical Trial. JAMA Ophthalmol. 2021 Jul 1;139(7):701-712. doi: 10.1001/jamaophthalmol.2021.0606. PMID 33784735

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Aflibercept: Aflibercept injection in study eye at randomization and at visits at 1, 2, and 4 months and then every 4 months thereafter. More frequent aflibercept may be given if center-involved diabetic macular edema or proliferative diabetic retinopathy develops and deferred laser may subsequently be added to intravitreal aflibercept if certain criteria are met.
  Prompt aflibercept: Intravitreal injection of 2.0mg aflibercept is performed on the day of randomization and visits at 1, 2, and 4 months and then every 4 months thereafter.
  Deferred laser: Laser (either focal/grid laser for diabetic macular edema or panretinal photocoagulation for proliferative diabetic retinopathy) is added following initiation of anti-vascular endothelial growth factor injections for center-involved diabetic macular edema or proliferative diabetic retinopathy only if certain criteria are met
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once proliferative diabetic retinopathy or center-involved diabetic macular edema develops and then up to every 4 weeks using defined treatment criteria.
- Sham: Sham injection in study eye at randomization and at visits at 1, 2, and 4 months and then every 4 months thereafter. Deferred aflibercept may be given if center-involved diabetic macular edema or proliferative diabetic retinopathy develops and deferred laser may subsequently be added to intravitreal aflibercept if certain criteria are met.
  Prompt Sham: A sham injection (syringe without a needle pressed against the injection site) is performed on the day of randomization and visits at 1, 2, and 4 months and then every 4 months thereafter.
  Deferred laser: Laser (either focal/grid laser for diabetic macular edema or panretinal photocoagulation for proliferative diabetic retinopathy) is added following initiation of anti-vascular endothelial growth factor injections for center-involved diabetic macular edema or proliferative diabetic retinopathy only if certain criteria are met
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once proliferative diabetic retinopathy or center-involved diabetic macular edema develops and then up to every 4 weeks using defined treatment criteria.
Period: Overall Study
Arm/Group | Aflibercept | Sham
Started | 200; 200 Eyes (Number of Eyes) | 199; 199 Eyes (Number of Eyes)
Completed | 160; 160 Eyes (Number of Eyes) | 167; 167 Eyes (Number of Eyes)
Not Completed | 40; 40 Eyes | 32; 32 Eyes
Not completed — Completed out of Window | 3 | 2
Not completed — Missed Visit | 5 | 2
Not completed — Lost to Follow-up | 12 | 7
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Death | 11 | 8

BASELINE CHARACTERISTICS:
Population: Units are in eyes. A participant could have 2 study eyes. For participants with two study eyes the participant was randomly assigned to receive sham in the eye with worse diabetic retinopathy and aflibercept in the other, or aflibercept in the eye with the worse diabetic retinopathy and sham in the other.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept | Sham | Total
Number analyzed (Participants) | 200 | 199 | 399
Number analyzed (Eyes) | 200 | 199 | 399
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [51 to 63] | 56 [48 to 62] | 57 [51 to 64]
Sex/Gender, Customized [Number; unit: Eyes]
  Female | 83 | 86 | 139
  Male | 117 | 113 | 189
Race/Ethnicity, Customized [Number; unit: Eyes]
  White | 92 | 86 | 178
  Hispanic or Latino | 62 | 67 | 129
  Black or African American | 29 | 32 | 61
  Asian | 10 | 9 | 19
  More than one race | 3 | 1 | 4
  Unknown | 2 | 3 | 5
  American Indian or Alaskan native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 1 | 2
Diabetes Type [Number; unit: Eyes]
  Type 1 | 12 | 23 | 35
  Type 2 | 188 | 176 | 364
Duration of Diabetes [Median (Inter-Quartile Range); unit: years] | 17 [10 to 22] | 16 [11 to 22] | 16 [10 to 22]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percent] — Hemoglobin A1c values were missing for 11 participants in the aflibercept group and 9 participants in the sham group
  Percent | 8.6 [7.1 to 10.0] | 8.3 [7.3 to 9.7] | 8.4 [7.2 to 9.9]
Mean arterial blood pressure [Median (Inter-Quartile Range); unit: mmHg] — Mean arterial blood pressure = (Systolic blood pressure + 2*Diastolic blood pressure) / 3
  mmHg | 100 [92 to 107] | 98 [91 to 106] | 99 [92 to 106]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 31 [28 to 37] | 31 [27 to 36] | 31 [28 to 36]
Prior myocardial infarction [Number; unit: Participant] | 16 | 19 | 35
Prior stroke [Number; unit: Participant] | 13 | 11 | 21
Pre-existing renal disease [Number; unit: Participant] | 6 | 6 | 11
Visual acuity [Mean (Inter-Quartile Range); unit: letter score] — Measure Description: Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  letter score | 88 [84 to 90] | 88 [85 to 91] | 88 [84 to 90]
Optical coherence tomography central subfield thickness [Median (Inter-Quartile Range); unit: Microns] — Heidelberg Spectralis machine equivalent. Spectralis = 40.78 + 0.95 × cirrus.
  Microns | 283 [264 to 300] | 283 [265 to 299] | 283 [264 to 299]
Diabetic retinopathy severity scale level [Number; unit: Eyes] — NPDR= Non-proliferative diabetic retinopathy
  Eyes
    Moderate NPDR (level 43) | 33 | 35 | 68
    Moderately severe NPDR (level 47A) | 65 | 61 | 126
    Moderately severe NPDR (level 47B-D) | 54 | 55 | 109
    Severe NPDR (level 53) | 48 | 48 | 96
Intraocular pressure [Median (Inter-Quartile Range); unit: mmHg] | 15 [13 to 17] | 15 [13 to 17] | 15 [13 to 17]
Lens status [Number; unit: Eyes]
  Posterior chamber Intraocular lens | 34 | 32 | 66
  Phakic | 166 | 167 | 333
Non-central diabetic macular edema [Number; unit: Eyes] — At least 2 noncentral macular subfields with optical coherence tomography (OCT) thickness above threshold (average normal + 2 SD) or at least 1 noncentral macular subfield with OCT thickness at least 15 μm above threshold (average normal + 2 SD). Population: Missing for 12 eyes in the aflibercept group and 4 eyes in the sham group
  Eyes
    number analyzed (Participants) | 188 | 195 | 383
    (all) | 75 | 83 | 158
Prior anti-vascular endothelial growth factor therapy for diabetic macular edema [Number; unit: Eyes] | 8 | 5 | 13
Prior focal or grid laser for diabetic macular edema [Number; unit: Eyes] | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Development of PDR and/or DME (Whichever Came First)
Description: CI-DME = center-involved diabetic macular edema, PDR = proliferative diabetic macular edema. First development of criteria meeting end point. Eyes that met any criteria are then censored from contributing to the next criteria. Eyes that did not meet the outcome were censored at the time of the last completed visit. Each outcome appears only once under "First PDR and/or DME criteria met." Outcomes appear under "Development of PDR" if PDR developed at any time in the study (regardless of if or when DME developed) and outcomes appear under "Development of DME" if DME developed at any time in the study (regardless of if or when PDR developed)
Time Frame: 2 years
Population: as for baseline characteristics
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept | Sham
Number analyzed (Participants) | 200 | 199
Number analyzed (Eyes) | 200 | 199
Eyes | 27 | 75

2. Primary Outcome: Change in Visual Acuity From Baseline
Description: Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Aflibercept | Sham
Number analyzed (Participants) | 160 | 166
Number analyzed (Eyes) | 160 | 166
Letter Score | -0.9 (5.8) | -2.0 (6.1)

3. Secondary Outcome: Change in Visual Acuity From Baseline
Description: as for outcome 2
Time Frame: 4 years
Population: Includes only eyes that completed the 4-year visit.
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Aflibercept | Sham
Number analyzed (Participants) | 137 | 134
Number analyzed (Eyes) | 137 | 134
Letter Score | -2.7 (6.5) | -2.4 (5.8)

4. Secondary Outcome: Development of PDR and/or DME (Whichever Came First)
Description: as for outcome 1
Time Frame: 4 years
Population: as for baseline characteristics
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Aflibercept | Sham
Number analyzed (Participants) | 200 | 199
Number analyzed (Eyes) | 200 | 199
Eyes | 54 | 97

ADVERSE EVENTS:
Time Frame: 2 Years
Description: To get the total number of participant/eyes in each treatment group add the unilateral and bilateral participants together:
  Unilateral Aflibercept = 129 Total aflibercept = unilateral aflibercept + bilateral = 129 + 71 = 200
  Unilateral sham = 128 total sham = unilateral sham + bilateral = 128 + 71 = 199
Groups:
- Bilateral Participants: Participants with one eye enrolled in each arm of the study.
Arm/Group | Aflibercept | Sham | Bilateral Participants
All-Cause Mortality (participants affected / at risk) | 9/129 | 10/128 | 5/71
Serious Adverse Events (participants affected / at risk) | 52/129 | 50/128 | 24/71
Other Adverse Events (participants affected / at risk) | 116/129 | 112/128 | 62/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=129) | Sham (N=128) | Bilateral Participants (N=71)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
AFib (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 6 (8) | 6 (8) | 2 (5)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Endocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5) | 6 (6) | 3 (3)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperglycemia (Endocrine disorders) | 1 (1) | 2 (2) | 2 (2)
Hyperglycemic hyperosmolar nonketotic syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Colitis collagenous (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
esophagus ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Death (General disorders) | 2 (2) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 0 (0)
Swelling of feet (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Helicobacter pylori infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Infection (chronic) of amputation stump (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MRSA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Septicemia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Staphylococcal infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Leg injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Charcot arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fractured ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Tendon disorder NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer (NOS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Desmoplastic small round cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Anoxic brain damage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage brain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurologic disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral neuropathy NOS (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
End stage renal disease (ESRD) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Kidney function abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Cellulitis of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bypass surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Feeding tube insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Embolism - blood clot (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension worsened (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Stroke (cerebrovascular accident) (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Stroke - Haemorrhagic (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischemic attacks (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=129) | Sham (N=128) | Bilateral Participants (N=71)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4) | 0 (0)
Anemia, unspecified (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Fluid in middle ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus poor control (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Graves' disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
Loss of control of blood sugar (Endocrine disorders) | 3 (3) | 2 (2) | 2 (2)
Thyroid nodule (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of diabetes (Endocrine disorders) | 5 (5) | 4 (4) | 3 (3)
Abnormal vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic conjunctivitis (Eye disorders) | 2 (2) | 1 (1) | 1 (2)
Anatomical narrow angle borderline glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anterior chamber angle neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anterior membrane dystrophy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Atrophy of macula (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (eyelid irritation) (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Blepharo conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 8 (8) | 7 (8) | 7 (16)
Blurry vision (Eye disorders) | 1 (1) | 3 (3) | 7 (9)
Burning eyes (Eye disorders) | 1 (1) | 1 (1) | 2 (4)
Cataract (Eye disorders) | 23 (24) | 26 (27) | 17 (26)
Cataract cortical (Eye disorders) | 5 (6) | 2 (2) | 2 (2)
Cataract subcapsular (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cloudy vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival cyst (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival injection (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1) | 1 (2)
Corneal abrasion (Eye disorders) | 6 (6) | 3 (4) | 2 (2)
Corneal disorder (NOS) (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal guttata (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal haze (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cortical spoking (Eye disorders) | 1 (1) | 3 (3) | 2 (3)
Cotton wool spots (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Cystoid macular edema (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic macular edema (Eye disorders) | 7 (7) | 14 (15) | 6 (7)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Disc neovascularization (Eye disorders) | 2 (2) | 3 (3) | 2 (2)
Distorted vision (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Dot hemorrhages (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Double vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 10 (11) | 9 (9) | 9 (12)
Epiretinal membrane (Eye disorders) | 3 (3) | 3 (3) | 2 (2)
Episcleritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye ache (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 6 (8) | 3 (6)
Eye itching (Eye disorders) | 2 (2) | 3 (3) | 3 (5)
Eye pain (Eye disorders) | 5 (5) | 6 (7) | 5 (8)
Eye strain (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Eye tearing (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Eye tired (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Eyelid edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid twitching (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 19 (19) | 6 (8) | 7 (9)
Fog in front of eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Glare (Eye disorders) | 1 (1) | 1 (1) | 1 (2)
Glaucoma (Eye disorders) | 2 (2) | 2 (2) | 1 (2)
Hazy vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hollenhorst plaque (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopyon (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraretinal microvascular abnormalities (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Iris neovascularization (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iritis (anterior uveitis, iridocyclitis) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemia retinal (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Ischemic optic neuropathy (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Keratopathy NOS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lid papilloma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular cyst (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular cyst, hole, or pseudohole of retina (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Macular edema (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Macular hole (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular ischemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Macular puckering (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Meibomian gland obstruction (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Near vision disturbance (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Nuclear sclerosis (Eye disorders) | 4 (4) | 5 (5) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 3 (3)
Optic nerve pallor (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 2 (2) | 1 (2)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Posterior capsule opacification (Eye disorders) | 6 (6) | 5 (5) | 2 (4)
Posterior subcapsular cataract (Eye disorders) | 10 (11) | 6 (6) | 4 (5)
Posterior vitreous detachment (Eye disorders) | 5 (5) | 2 (2) | 5 (5)
Preglaucoma, unspecified (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Preproliferative diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Preretinal hemorrhage (Eye disorders) | 0 (0) | 5 (5) | 1 (2)
Proliferative diabetic retinopathy (Eye disorders) | 2 (2) | 9 (9) | 7 (7)
Ptosis (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Punctate epithelial erosion (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Red eye (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Retinal disorder NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal exudates (Eye disorders) | 0 (0) | 3 (4) | 2 (2)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal neovascularization (Eye disorders) | 4 (5) | 5 (5) | 4 (4)
Retinal nonperfusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal vein disorder NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal vessel avulsion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinoschisis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Sensitivity to light (photophobia) (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Silicone oil droplets (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Spots before eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Stye (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
Subconjunctival hemorrhage (Eye disorders) | 8 (17) | 6 (6) | 3 (3)
Subconjunctival/conjunctival hemorrhage (Eye disorders) | 2 (2) | 1 (1) | 1 (2)
Subhyaloid hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial punctate keratitis (Eye disorders) | 0 (0) | 4 (4) | 3 (6)
Traction retinal detachment (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vision decreased (Eye disorders) | 4 (5) | 2 (2) | 2 (4)
Visual acuity decreased (Eye disorders) | 0 (0) | 3 (3) | 1 (2)
Visual disturbances (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual flashes (Eye disorders) | 0 (0) | 2 (2) | 2 (3)
Visual impairment transient (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreomacular traction syndrome (Eye disorders) | 1 (1) | 2 (4) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Vitreous floater (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Vitreous hemorrhage (Eye disorders) | 7 (9) | 18 (21) | 5 (7)
Watering eyes (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Acid reflux (oesophageal) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Anal irritation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bowel incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
External hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2)
Gastrointestinal stromal tumor (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Internal hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 0 (0)
Oral lesion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sessile colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomach virus (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Tooth abscess (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Tooth fracture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Catheter infection (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 2 (3) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1)
Fever (General disorders) | 4 (4) | 1 (1) | 1 (1)
General Swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 2 (3)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Leg edema (General disorders) | 3 (4) | 4 (4) | 1 (1)
Lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain NOS (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pain in face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pedal edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Swelling of feet (General disorders) | 1 (1) | 2 (2) | 1 (1)
Tiredness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy NOS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Gluten intolerance (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (3) | 2 (2) | 0 (0)
Systemic lupus erythematosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess NOS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Acute pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Helicobacter pylori infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected toe (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (4) | 2 (2) | 3 (3)
Infection NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (7) | 6 (6) | 3 (3)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MRSA (Infections and infestations) | 2 (4) | 2 (2) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection NOS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral syndrome (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Yeast infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bee sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bug bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (8) | 3 (4)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Laceration of leg (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spider bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Arteriogram (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine abnormal NOS (Investigations) | 0 (0) | 1 (1) | 0 (0)
Elevated liver enzymes (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated white cell count (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glucose high (Investigations) | 1 (1) | 0 (0) | 0 (0)
HbA1C increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate low (Investigations) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 2 (2) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Testosterone low (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Dyslipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Fluid overload - fluid volume increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesteremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Unintentional weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 1 (1)
Water retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 2 (2)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone spur (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Broken foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Broken wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Chest tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dislocated shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Fractured tailbone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fractured toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Frozen shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3)
Lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in heel (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Shoulder discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Sore tailbone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sprain of unspecified site of wrist (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sprains and strains of ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (3)
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast lump (benign) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Polyp of vocal cord or larynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Diabetic peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial droop (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fainting (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Head pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 8 (9) | 2 (6)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Numbness in feet (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Numbness in hand (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Post herpetic neuralgia (infection) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis of unspecified region (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Vasovagal attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mental state abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Azotemia prerenal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 6 (6) | 2 (2)
Chronic renal failure worsened (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
End stage renal disease (ESRD) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (blood in urine) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Kidney function abnormal (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (2)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 6 (10) | 7 (7) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urination frequency of (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal disorder NOS (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 2 (2)
Bronchitis asthmatic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Cold (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (5) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (6) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Streptococcal sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (7) | 1 (4)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister of foot and toe(s), without mention of infection (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of arm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatochalasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Ecchymosis - skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Epidermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythematous conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hair thinning (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Poison ivy rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Skin callus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Achilles tendon elongation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Atherectomy (Surgical and medical procedures) | 0 (0) | 1 (3) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Cataract extraction (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (2)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Dental implantation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Foot surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee surgery NOS (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 2 (2) | 1 (2) | 1 (2)
Toe amputation (Surgical and medical procedures) | 3 (3) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 3 (3) | 1 (1)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Atherosclerosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Embolism - blood clot (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 7 (7) | 5 (5) | 1 (1)
Hypertension worsened (Vascular disorders) | 9 (9) | 6 (7) | 6 (8)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose veins (Vascular disorders) | 0 (0) | 2 (3) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02634333/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02634333/SAP_001.pdf